CLINICAL TRIAL: NCT03726359
Title: Phase I TITE-CREM Dose Escalation Study of Fractionated Stereotactic Radiation Therapy (FSRT) in Unresected Brain Metastases
Brief Title: Phase I Study of Fractionated Stereotactic Radiation Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-8344
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fractionated Stereotactic Radiation Therapy (FSRT) (Experimental): This study is unique in that it employs a continuous reassessment methodology (CRM) to determine the Maximum Tolerated Dose. Information for the proper dose level for each subsequent patient enrolled will be determined based on DLTs from previous patients enrolled in the trial.
  Interventions: Radiation: Fractionated Stereotactic Radiation Therapy (FSRT)

INTERVENTIONS:
Radiation: Fractionated Stereotactic Radiation Therapy (FSRT) — Initial starting dose will be 7 Gy x5= 35 Gy delivered to the planning target volume (PTV). Radiotherapy will be delivered every other day so that the Stereotactic Body Radiation Therapy (SBRT) schedule is completed within 1.5-2 weeks.

SUMMARY:
There is a lack of prospective trial data and consensus guidelines describing the use of Fractionated Stereotactic Radiation Therapy (FSRT) in the treatment of brain metastases. There has been no prospective dose escalation study performed to date to determine the maximum tolerated dose (MTD) in patients treated with FSRT. Prescription doses in the series described above ranged from 18 Gy to 42 Gy, delivered in 3 to 12 fractions. The results of this study will be used to plan future Phase II/III studies to determine the efficacy of different dose fractionation schedules of FSRT. The investigator team thus proposes a Phase I study to determine the feasibility and safety of FSRT in patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of a non-hematological malignancy other than small cell lung cancer within 5 years of registration
* Intact (unresected) brain metastases measuring ≥3 cm and ≤ 6 cm in largest dimension on gadolinium contrast enhanced MRI obtained within 30 days prior to registration OR Surgically resected brain metastasis for which postoperative stereotactic radiotherapy is indicated, with expected target measuring ≥3 cm and ≤6 cm in largest dimension
* Prior Whole Brain Radiation Therapy (WBRT) is allowed
* Age ≥ 18 years
* Women of childbearing potential and male participants must practice adequate contraception
* History/Physical examination within 30 days prior to registration
* Life expectancy >3 months
* Patients are allowed to enroll if previously treated to other lesions with Stereotactic Radiosurgery (SRS)
* Patients with multiple lesions are allowed, as long there is one dominant lesion that will be treated with FSRT. Other lesions may be treated concurrently with SRS or FSRT at the discretion of the treating physician but will not contribute to the study endpoints

Exclusion Criteria:

* Patients with definitive leptomeningeal metastases, based on cerebrospinal fluid (CSF) examination
* Plan for chemotherapy or targeted agents during treatment. Hormonal therapy, immunotherapy targeting PD-1/PD-L1 axis, and bone supportive therapy may be continued during treatment
* Contraindication to enhanced MRI imaging such as implanted metal devices. However, patients with implanted devices which are MRI compatible are allowed
* Patients with measurable brain metastasis resulting from small cell lung cancer and germ cell malignancy
* Uncontrolled intercurrent illness such as congestive heart failure, unstable angina, cardiac arrhythmia, and uncontrolled seizure activity
* Previous treatment of the target lesion with radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within 1 year of initiation of treatment
  Determine the maximum tolerated dose (MTD) associated with a 20% dose limiting toxicity (DLT). DLT is defined as grade 3 or higher toxicities that occur within 1 year of treatment start and either possibly, probably, or definitively related to radiotherapy (RT).

SECONDARY OUTCOMES:
Response to Treatment | Up to 1 year following initiation of treatment
  Response to treatment will be assessed based on the percentage of patients who achieve either a complete response (CR), partial response (PR), or stable disease (SD), or progression (P) in response to FSRT treatment will be determined. Best response will be summarized. Response criteria will be assessed as follows
  Complete Response (CR): Defined as follow up imaging which shows that complete radiographic disappearance of brain metastasis. Partial Response (PR): Decrease of >50% in the size of each lesion radiographically, using perpendicular diameters Stable Disease (SD): 0 to 50% reduction in size of each lesion radiographically, using perpendicular diameters. Progression (P): Defined as > 25% increase in the size of each lesion or a new, non-contiguous lesion developed outside of the radiosurgical volume.

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin X, DeAngelis LM. Treatment of Brain Metastases. J Clin Oncol. 2015 Oct 20;33(30):3475-84. doi: 10.1200/JCO.2015.60.9503. Epub 2015 Aug 17. PMID 26282648
- [Background] Patchell RA, Tibbs PA, Walsh JW, Dempsey RJ, Maruyama Y, Kryscio RJ, Markesbery WR, Macdonald JS, Young B. A randomized trial of surgery in the treatment of single metastases to the brain. N Engl J Med. 1990 Feb 22;322(8):494-500. doi: 10.1056/NEJM199002223220802. PMID 2405271
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Li J, Bentzen SM, Renschler M, Mehta MP. Regression after whole-brain radiation therapy for brain metastases correlates with survival and improved neurocognitive function. J Clin Oncol. 2007 Apr 1;25(10):1260-6. doi: 10.1200/JCO.2006.09.2536. PMID 17401015
- [Background] Welzel G, Fleckenstein K, Schaefer J, Hermann B, Kraus-Tiefenbacher U, Mai SK, Wenz F. Memory function before and after whole brain radiotherapy in patients with and without brain metastases. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1311-8. doi: 10.1016/j.ijrobp.2008.03.009. Epub 2008 Apr 28. PMID 18448270
- [Background] Meyers CA, Smith JA, Bezjak A, Mehta MP, Liebmann J, Illidge T, Kunkler I, Caudrelier JM, Eisenberg PD, Meerwaldt J, Siemers R, Carrie C, Gaspar LE, Curran W, Phan SC, Miller RA, Renschler MF. Neurocognitive function and progression in patients with brain metastases treated with whole-brain radiation and motexafin gadolinium: results of a randomized phase III trial. J Clin Oncol. 2004 Jan 1;22(1):157-65. doi: 10.1200/JCO.2004.05.128. PMID 14701778
- [Background] Brown PD, Pugh S, Laack NN, Wefel JS, Khuntia D, Meyers C, Choucair A, Fox S, Suh JH, Roberge D, Kavadi V, Bentzen SM, Mehta MP, Watkins-Bruner D; Radiation Therapy Oncology Group (RTOG). Memantine for the prevention of cognitive dysfunction in patients receiving whole-brain radiotherapy: a randomized, double-blind, placebo-controlled trial. Neuro Oncol. 2013 Oct;15(10):1429-37. doi: 10.1093/neuonc/not114. Epub 2013 Aug 16. PMID 23956241
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Kondziolka D, Patel A, Lunsford LD, Kassam A, Flickinger JC. Stereotactic radiosurgery plus whole brain radiotherapy versus radiotherapy alone for patients with multiple brain metastases. Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):427-34. doi: 10.1016/s0360-3016(99)00198-4. PMID 10487566
- [Background] Aoyama H, Tago M, Shirato H; Japanese Radiation Oncology Study Group 99-1 (JROSG 99-1) Investigators. Stereotactic Radiosurgery With or Without Whole-Brain Radiotherapy for Brain Metastases: Secondary Analysis of the JROSG 99-1 Randomized Clinical Trial. JAMA Oncol. 2015 Jul;1(4):457-64. doi: 10.1001/jamaoncol.2015.1145. PMID 26181254
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Shaw E, Scott C, Souhami L, Dinapoli R, Kline R, Loeffler J, Farnan N. Single dose radiosurgical treatment of recurrent previously irradiated primary brain tumors and brain metastases: final report of RTOG protocol 90-05. Int J Radiat Oncol Biol Phys. 2000 May 1;47(2):291-8. doi: 10.1016/s0360-3016(99)00507-6. PMID 10802351
- [Background] Minniti G, Clarke E, Lanzetta G, Osti MF, Trasimeni G, Bozzao A, Romano A, Enrici RM. Stereotactic radiosurgery for brain metastases: analysis of outcome and risk of brain radionecrosis. Radiat Oncol. 2011 May 15;6:48. doi: 10.1186/1748-717X-6-48. PMID 21575163
- [Background] Vogelbaum MA, Angelov L, Lee SY, Li L, Barnett GH, Suh JH. Local control of brain metastases by stereotactic radiosurgery in relation to dose to the tumor margin. J Neurosurg. 2006 Jun;104(6):907-12. doi: 10.3171/jns.2006.104.6.907. PMID 16776334
- [Background] Yang HC, Kano H, Lunsford LD, Niranjan A, Flickinger JC, Kondziolka D. What factors predict the response of larger brain metastases to radiosurgery? Neurosurgery. 2011 Mar;68(3):682-90; discussion 690. doi: 10.1227/NEU.0b013e318207a58b. PMID 21311296
- [Background] Blonigen BJ, Steinmetz RD, Levin L, Lamba MA, Warnick RE, Breneman JC. Irradiated volume as a predictor of brain radionecrosis after linear accelerator stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):996-1001. doi: 10.1016/j.ijrobp.2009.06.006. Epub 2009 Sep 23. PMID 19783374
- [Background] Aoyama H, Shirato H, Onimaru R, Kagei K, Ikeda J, Ishii N, Sawamura Y, Miyasaka K. Hypofractionated stereotactic radiotherapy alone without whole-brain irradiation for patients with solitary and oligo brain metastasis using noninvasive fixation of the skull. Int J Radiat Oncol Biol Phys. 2003 Jul 1;56(3):793-800. doi: 10.1016/s0360-3016(03)00014-2. PMID 12788187
- [Background] Eaton BR, Gebhardt B, Prabhu R, Shu HK, Curran WJ Jr, Crocker I. Hypofractionated radiosurgery for intact or resected brain metastases: defining the optimal dose and fractionation. Radiat Oncol. 2013 Jun 7;8:135. doi: 10.1186/1748-717X-8-135. PMID 23759065
- [Background] Ernst-Stecken A, Ganslandt O, Lambrecht U, Sauer R, Grabenbauer G. Phase II trial of hypofractionated stereotactic radiotherapy for brain metastases: results and toxicity. Radiother Oncol. 2006 Oct;81(1):18-24. doi: 10.1016/j.radonc.2006.08.024. Epub 2006 Sep 15. PMID 16978720
- [Background] Fahrig A, Ganslandt O, Lambrecht U, Grabenbauer G, Kleinert G, Sauer R, Hamm K. Hypofractionated stereotactic radiotherapy for brain metastases--results from three different dose concepts. Strahlenther Onkol. 2007 Nov;183(11):625-30. doi: 10.1007/s00066-007-1714-1. PMID 17960338
- [Background] Feuvret L, Vinchon S, Martin V, Lamproglou I, Halley A, Calugaru V, Chea M, Valery CA, Simon JM, Mazeron JJ. Stereotactic radiotherapy for large solitary brain metastases. Cancer Radiother. 2014 Mar;18(2):97-106. doi: 10.1016/j.canrad.2013.12.003. Epub 2014 Jan 14. PMID 24439342
- [Background] Rajakesari S, Arvold ND, Jimenez RB, Christianson LW, Horvath MC, Claus EB, Golby AJ, Johnson MD, Dunn IF, Lee EQ, Lin NU, Friesen S, Mannarino EG, Wagar M, Hacker FL, Weiss SE, Alexander BM. Local control after fractionated stereotactic radiation therapy for brain metastases. J Neurooncol. 2014 Nov;120(2):339-46. doi: 10.1007/s11060-014-1556-5. Epub 2014 Jul 25. PMID 25059451
- [Background] Jiang XS, Xiao JP, Zhang Y, Xu YJ, Li XP, Chen XJ, Huang XD, Yi JL, Gao L, Li YX. Hypofractionated stereotactic radiotherapy for brain metastases larger than three centimeters. Radiat Oncol. 2012 Mar 19;7:36. doi: 10.1186/1748-717X-7-36. PMID 22429918
- [Background] Kim YJ, Cho KH, Kim JY, Lim YK, Min HS, Lee SH, Kim HJ, Gwak HS, Yoo H, Lee SH. Single-dose versus fractionated stereotactic radiotherapy for brain metastases. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):483-9. doi: 10.1016/j.ijrobp.2010.05.033. Epub 2010 Aug 26. PMID 20800386
- [Background] Kwon AK, Dibiase SJ, Wang B, Hughes SL, Milcarek B, Zhu Y. Hypofractionated stereotactic radiotherapy for the treatment of brain metastases. Cancer. 2009 Feb 15;115(4):890-8. doi: 10.1002/cncr.24082. PMID 19132728
- [Background] Lederman G, Wronski M, Fine M. Fractionated radiosurgery for brain metastases in 43 patients with breast carcinoma. Breast Cancer Res Treat. 2001 Jan;65(2):145-54. doi: 10.1023/a:1006490200335. PMID 11261830
- [Background] Ma LH, Li G, Zhang HW, Wang ZY, Dang J, Zhang S, Yao L, Zhang XM. Hypofractionated stereotactic radiotherapy with or without whole-brain radiotherapy for patients with newly diagnosed brain metastases from non-small cell lung cancer. J Neurosurg. 2012 Dec;117 Suppl:49-56. doi: 10.3171/2012.7.GKS121071. PMID 23205789
- [Background] Minniti G, D'Angelillo RM, Scaringi C, Trodella LE, Clarke E, Matteucci P, Osti MF, Ramella S, Enrici RM, Trodella L. Fractionated stereotactic radiosurgery for patients with brain metastases. J Neurooncol. 2014 Apr;117(2):295-301. doi: 10.1007/s11060-014-1388-3. Epub 2014 Feb 1. PMID 24488446
- [Background] Wiggenraad R, Verbeek-de Kanter A, Kal HB, Taphoorn M, Vissers T, Struikmans H. Dose-effect relation in stereotactic radiotherapy for brain metastases. A systematic review. Radiother Oncol. 2011 Mar;98(3):292-7. doi: 10.1016/j.radonc.2011.01.011. PMID 21316787
- [Background] Baliga S, Garg MK, Fox J, Kalnicki S, Lasala PA, Welch MR, Tome WA, Ohri N. Fractionated stereotactic radiation therapy for brain metastases: a systematic review with tumour control probability modelling. Br J Radiol. 2017 Feb;90(1070):20160666. doi: 10.1259/bjr.20160666. Epub 2016 Dec 12. PMID 27936894